CLINICAL TRIAL: NCT00551343
Title: Contribution of a GLP-1 Agonist to Appetite Regulation, Metabolism and Body Composition in Subjects With Prader-Willi Syndrome.
Brief Title: Gut Derived Hormones, Body Composition and Metabolism in Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H07/045; X07-0178
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2007-10

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PWS (Other)
  Interventions: Drug: Exenatide
- Controls (Other)
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 10ug Exenatide single s.c. injection

SUMMARY:
The purpose of this study is to investigate the effects of a GLP-1 agonist on satiety hormones in patients with Prader-Willi Syndrome (genetic defect causing obesity).

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is the most frequent known genetic disorder of obesity. Hyperphagia is the main barrier to independent living in adults with PWS, and hitherto behavioural restraints and environmental modification are the only effective management measure. The emerging costs for professional care are immense. Thus, there is an urgent need for treatment which reduce appetite and food intake in this patient group. Agonists of the gut derived hormone GLP-1 which reduces food intake and causes weight loss due to slowed gastric emptying and through direct central effects. The aim of this pilot drug trial is to analyse the effect of a GLP-1 agonist on appetite regulating hormones, insulin secretion and energy expenditure before and after a meal.

ELIGIBILITY:
Inclusion Criteria:

* see below

Exclusion Criteria:

* Diabetes mellitus, acute infections

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
satiety hormones | 1 day

SECONDARY OUTCOMES:
appetite (visual analogue scale) insulin secretion | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lesley V Campbell, Prof, Principal Investigator — Garvan Institute of Medical Research
Locations (1):
- Garvan Institute of Medical Research, Sydney, New South Wales, Australia